CLINICAL TRIAL: NCT00863538
Title: An Open-label, Phase II Study of KPS-0373 in Patients With SCD
Brief Title: Phase II Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPS1201
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration; Thyrotropin-Releasing Hormone (TRH); SCD
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: KPS-0373

INTERVENTIONS:
Drug: KPS-0373

SUMMARY:
To evaluate the efficacy, safety and pharmacokinetics profile of KPS-0373 in patients with SCD

ELIGIBILITY:
Inclusion Criteria:

* SCD with mild to moderate ataxia

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA), ADL(Flow-FIM), Patient Improvement Impression | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (3):
- Japan (3):
  - Japan, Hokkaido Region
  - Japan, Kansai Region
  - Japan, Kanto Region